CLINICAL TRIAL: NCT04523649
Title: Protocol for Rationale and Design of Home-Based SolUtion for Remote Atrial Fibrillation Screening to PrevenT RecUrrence StrOke (HUA-TUO AF Trial): A Randomized Open-label Study
Brief Title: Home-Based SolUtion for Remote Atrial Fibrillation Screening to PrevenT RecUrrence StrOke (HUA-TUO AF Trial)
Acronym: HUA-TUO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HUA-TUO
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Stroke, Cardiovascular
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centered, randomized controlled, parallel-group study
Who Masked: Outcomes Assessor
Masking Description: Independent research officers and data staff responsible for data entry will be blinded from randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based atrial fibrillation screening group (Experimental): Patients in this group will be given a handheld single lead ECG recorder (Comfit Healthcare Devices Limited, Hong Kong SAR, China) and a patient-facing smartphone application specially designed for the study, and they will be requested to record daily ECG and certain vital measurement.
  Interventions: Device: Remote atrial fibrillation screening with handheld single lead ECG recorder
- Control group (No Intervention): Conventional medical care

INTERVENTIONS:
Device: Remote atrial fibrillation screening with handheld single lead ECG recorder — Patients in this group will be given a handheld single lead ECG recorder (Comfit Healthcare Devices Limited, Hong Kong SAR, China) and a patient-facing smartphone application specially designed for the study, and they will be requested to record daily ECG and certain vital measurement.
  Arms: Home-based atrial fibrillation screening group

SUMMARY:
Stroke remains the leading cause of mortality and morbidity worldwide. Patients surviving the first ever stroke remain at high risk of stroke recurrence. While the cause of stroke recurrence is multifactional, atrial fibrillation (AF) has been recognized as one of the most important factors for stroke recurrence. Despite the fact that AF related stroke is highly preventable with long-term oral anticoagulation therapy particularly the non-vitamin K oral anticoagulants (NOAC), the arrhythmia is often not diagnosed until stroke recurrence due to its paroxysmal and asymptomatic nature.

Diagnosing AF before stroke recurrence has been recognized as one of the most important objectives for stroke management. Strategies to detection AF in stroke survivors have been recommended including 7-day or 14-day Holter monitoring at the early post-stroke period. There's also study trial exploring the clinical application of insertable cardiac monitor to detect AF in patients with recent cryptogenic stroke.

In the past decade, advance in ECG technology has made possible to record ECG using handheld smartphone accessory devices in household setting. Together with the rapid developing artificial intelligence-based ECG diagnosis and mobile communication, it is possible to remotely monitor hundreds of thousand ECGs from patients at risk of AF. Few randomized trials have assessed the effectiveness of handheld ECG recording device for AF detection in patients with history of stroke. Here we test the hypothesis that long-term home-based ECG monitoring will be more sensitive than standard care in detecting AF in patients with history of stroke but no documented AF for 24 months. Secondarily, we will investigate whether early detection of AF might confer a benefit on longer-term clinical outcomes.

DETAILED DESCRIPTION:
The trial will primarily be conducted in Hong Kong SAR, Macau SAR, and mainland China. It is a prospective, multi-centered, randomized controlled, parallel-group study to compare the time to detect AF with portable handheld single lead ECG recorder versus conventional care in patients with history of ischemic stroke without documented AF. Patients will be randomly assigned in a 1:1 ratio to Home-based AF screening group and Control group.

The home-based AF screening system comprises (1) a handheld single lead electrocardiogram (ECG) recorder (Comfit Healthcare Devices Limited, Hong Kong SAR, China), and (2) a patient-facing smartphone application specially designed for the study. Patients randomized to the home-based AF group will be instructed to record a 30-second single lead ECG using the handheld ECG device every morning or when symptomatic. In addition, all study participants will be instructed to measure and report their blood pressures in the morning and evening through the patient-facing smartphone application. In addition, all study participants will be encouraged to input their routine blood tests from the public hospitals through the smartphone application.

All remotely obtained data will be automatically transmitted in real-time through the study smartphone application to a secured cloud hosting and displayed to display on a web-based dashboard at the clinicians' offices for review. All ECG recordings will be analyzed using an artificial intelligence based diagnosed system. When a diagnosis of AF is made with the system, the patients will be called back for a formal cardiology consultation and standard 12-lead ECG to confirm the diagnosis within 1 week. This will be followed by echocardiogram and blood tests to determine the possible options of long-term anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* history of ischemic stroke within 5 years
* voluntarily agrees to participate by providing written informed consent

Exclusion Criteria:

* previously documented AF and/or atrial flutter
* long-term anticoagulation therapy
* short life expectance (< 1year) due to concomitant medical condition(s)
* cardiac implantable electronic device
* inability or refusal to provide inform consent
* lack of skills in operating simple electronic devices
* unavailability of a mobile network service in the place of residence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1740 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
First detection of AF | 2 years
  First detection of AF by the handheld ECG, defined as an episode of irregular heart rhythm, without detectable P waves, lasting more than 30 seconds

SECONDARY OUTCOMES:
Recurrent stroke | 2 years
  Existence of subsequent stroke after joining the study
Transient ischemic attack (TIA) | 2 years
  Existence of subsequent TIA after joining the study
Initiation of long-term anticoagulation therapy | 2 years
  Initiation of long-term anticoagulation therapy after joining the study for any medical purposes
Hospitalization of heart failure | 2 years
  First hospitalization of heart failure after joining the study
Cardiovascular death | 2 years
  Death due to cardiovascular reasons after joining the study
All-cause death | 2 years
  Death due to all causes after joining the study

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Wah David Siu, Prof, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Dataset used during the study will be available from the corresponding author on reasonable request from date of publication for 2 years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Dataset used during the study will be available from the corresponding author on reasonable request from date of publication for 2 years.
Access Criteria: Dataset used during the study will be available from the corresponding author on reasonable request from date of publication for 2 years.

REFERENCES:
- [Derived] Wong CK, Hai JJ, Lau YM, Zhou M, Lui HW, Lau KK, Chan KH, Mok TM, Liu Y, Feng Y, Tan N, Tam WC, Tam KC, Feng X, Zuo ML, Yin LX, Tan J, Zhang WJ, Jiang X, Huang X, Ye J, Liang Y, Jiang W, Lei Z, Huang D, Yue WS, Tan G, Yan BP, Evora MA, Chen JY, Siu CW. Protocol for Home-Based Solution for Remote Atrial Fibrillation Screening to Prevent Recurrence Stroke (HUA-TUO AF Trial): a randomised controlled trial. BMJ Open. 2022 Jul 15;12(7):e053466. doi: 10.1136/bmjopen-2021-053466. PMID 35840293